CLINICAL TRIAL: NCT03580213
Title: Hand Therapy or Not Following Collagenase Treatment for Dupuytren's Contracture?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/613
Record Dates: First submitted 2018-04-10; First posted 2018-07-09 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-03

CONDITIONS: Dupuytren Disease of Palm and Finger, With Contracture
Keywords: Occupational Therapy; Physical Therapy; Hand Therapy; ADL; COPM; URAM; ROM; Hand exercise; Scar; Oedema; Splint; Orthosis
MeSH Terms: conditions — Dupuytren Contracture; Cicatrix; Edema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hand therapy MCPJ affected (Experimental): 40 participants With Dupuytren's contracture with only the Metacarpophalangeal joints affected, receiving hand therapy after collagenase injection and extension treatment.
  Hand therapy: edema control, wound and scar treatment, splinting, exercises for hand, exercise through activities of daily living.
  Interventions: Other: Hand therapy MCPJ affected
- Hand therapy PIPJ affected (Experimental): 40 participants With Dupuytren's contracture with the proximal interphalangeal joint involved, receiving hand therapy after collagenase injection and extension treatment.
  Hand therapy: edema control, wound and scar treatment, splinting, exercises for hand, exercise through activities of daily living. Possible additional splint and exercises specifically for the PIPJ extension.
  Interventions: Other: Hand therapy PIPJ affected
- Control group MCPJ affected (No Intervention): 40 participants With Dupuytren's contracture with only the Metacarpophalangeal joints affected.
  No treatment after the collagenase injection and extension treatment.
- Control group PIPJ affected (No Intervention): 40 participants With Dupuytren's contracture with only the Metacarpophalangeal joints affected.
  No treatment after the collagenase injection and extension treatment.

INTERVENTIONS:
Other: Hand therapy MCPJ affected — Prevention of oedema, treatment of scar, splinting to maintain or improve extension, exercises, activity of daily living as exercise. Instructions, demonstration and advices.
  Arms: Hand therapy MCPJ affected
Other: Hand therapy PIPJ affected — Prevention of oedema, treatment of scar, splinting to maintain or improve extension, exercises, activity of daily living as exercise. Instructions, demonstration and advices. Possible additional splint and exercises specifically for the PIPJ extension.
  Arms: Hand therapy PIPJ affected

SUMMARY:
This study evaluates if hand therapy have an impact on the patients' preformance of and satisfaction with everyday activities or not following collagenase injection treatment for Dupuytren's contracture. Differences on this between patients with contracted proximal interphalangeal joint(s) and patients with affected metacarpophalangeal joint(s) only, will also be investigated. Two equal sized groups will either receive hand therapy or no treatment following the injection and extension procedure.

DETAILED DESCRIPTION:
Today it varies if patients with collagenase treated Dupuytren's contracture (DC) are referred to hand therapy or not. No studies are found looking at the effect of therapy following collagenase treatment compared to no therapy.

The main purpose of the study is to find if hand therapy improves patients' performance of and satisfaction with everyday activities or not, one year after collagenase treatment for DC. Differences on this between patients with contracted proximal interphalangeal joint(s) (PIPJ) and patients with affected metacarpophalangeal joint(s) (MCPJ) only, will also be investigated.

A Norwegian randomised controlled trial will be conducted with two parallel intervention groups in a pre-test - post-test design. Hand therapy includes oedema control, scar management, night-time splinting, movement exercises and use of everyday activities as therapy. Additional individualised therapy will be provided if needed. Test times are right before, straight after, six weeks, four months and one year after collagenase treatment. Sample size needed is 160 participants. Appropriate methods of statistical analysis will be used.

Discussion Research on DC is challenging as the clinical picture is heterogeneous, no cure exists and no agreement on who should receive collagenase treatment. Hand therapy in the study will be individualised and not equal for every patient.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with collagenase injection and extension procedure for Dupuytren's contracture

Exclusion Criteria:

* earlier injury or treatment for Dupuytren's contracture in the same finger
* patients not capable of following a therapy program
* before randomisation: infection or an allergic reaction to the drug or Complex regional pain syndrome arising
* earlier participation in the same study makes the participant not eligible to be included once more when treated in the other hand.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) change from baseline to 6 weeks, from baseline to 4 months and to 1 year. | change from baseline to 6 weeks, baseline to 4 months and to 1 year.
  An individualized, client-centred outcome measure. COPM is an evidence-based outcome measure designed to capture a patient's self-perception of performance in everyday living, over time.

SECONDARY OUTCOMES:
Change on Unité Rhumatoloique des Affections de la Main (URAM) scale results from baseline to 6 weeks, from baseline to 4 months and to 1 year. | Change from Baseline to 6 weeks, from baseline to 4 months and to 1 year
  URAM, the Norwegian translation will be used. The scale evaluates the patients ability to perform 9 specific daily activities, which the patient are asked to score. The values are 6 ranges of difficulty: from no difficulties with doing the activity (score 0) to impossible to do (score 5). The possible total score ranges from 0 to 45, where 45 is the worse case.
Change on Range of motion (ROM) from baseline to 6 weeks, from baseline to 4 months and to 1 year. | Change from Baseline to 6 weeks, from baseline to 4 months and to 1 year
  Each affected joint will be measured for movement in extension and flexion with a goniometer.
Change on Visual Analogue Scale of pain (VAS) from baseline to 6 weeks, from baseline to 4 months and to 1 year. | Change from Baseline to 6 weeksfrom baseline to 4 months and to 1 year
  Visual analogue scale of pain. The patient scores from 0-10cm how much pain they have had the last week. No pain is scored 0 and worse pain is 10.
Change in grip force from baseline to 6 weeks, from baseline to 4 months and to 1 year. | Change from Baseline to 6 weeks from baseline to 4 months and to 1 year
  Jamar dynamometer

OTHER OUTCOMES:
Change in sensitivity to cold from baseline to 6 weeks, from baseline to 4 months and to 1 year. | Change from Baseline to 6 weeks from baseline to 4 months and to 1 year
  yes/no
Change in sick-leave status from baseline to 6 weeks, from baseline to 4 months and to 1 year. | Change from Baseline to 6 weeks from baseline to 4 months and to 1 year
  yes/no
Patient liability | Measured at 1 year from baseline
  Did the patient do as the protocol for therapy instructed? yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Terese Aglen, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aglen T, Matre KH, Lind C, Selles RW, Assmus J, Taule T. Hand therapy or not following collagenase treatment for Dupuytren's contracture? Protocol for a randomised controlled trial. BMC Musculoskelet Disord. 2019 Aug 28;20(1):387. doi: 10.1186/s12891-019-2712-z. PMID 31455312